CLINICAL TRIAL: NCT03076125
Title: Stroke Counseling for Risk Reduction in Young Adult African Americans
Brief Title: Stroke COunseling for Risk REduction
Acronym: SCORRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Dawn Aycock, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K01NR015494 (NIH)
Record Dates: First submitted 2017-03-05; First posted 2017-03-10 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: Primary Stroke Prevention, Risk Factors for Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: randomized controlled two-group pre-post test design
Who Masked: Participant, Outcomes Assessor
Masking Description: data collectors conducting post-intervention and 8-week follow up are blinded to participant treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCORRE group (Experimental): Stroke risk factor brochure, stroke champions video, counseling on accuracy of perceived stroke risk and strategies to reduce stroke risk, weekly motivational health behavior tips (for physical activity, diet, or smoking cessation) text messages for 8 weeks.
  Interventions: Behavioral: SCORRE
- Attention Control Group (Sham Comparator): Sexual health education brochure and Safe in the City video, weekly sexual health tips text messages for 8 weeks.
  Interventions: Behavioral: Attention-Control Activity

INTERVENTIONS:
Behavioral: SCORRE — 3 components based on the Health Belief Model
  Arms: SCORRE group
Behavioral: Attention-Control Activity — sexual health education
  Arms: Attention Control Group

SUMMARY:
The purpose of this study is to test the efficacy of the Stroke Counseling for Risk Reduction (SCORRE) intervention in increasing accuracy of perceived stroke risk and promoting lifestyle behavior change to reduce stroke risk in young adult African Americans.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American/Black
* age 20-35 years
* able to complete two study visits lasing 1 1/2- 2 hours and a brief daily diary for 8 weeks
* has a cell phone or email address to receive weekly reminders and tips
* has at least one modifiable risk factor for stroke identified during study visit one screening

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of perceived stroke risk | immediately post-intervention
  Comparison of perceived versus actual stroke risk
Targeted health behaviors | 8 weeks
  Improvements in targeted health behavior (physical activity, diet, or cigarette smoking)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No